CLINICAL TRIAL: NCT01818882
Title: Evaluation of the Diagnostic Value of Portable Ultrasound for Dyspneic Patient Support in the Emergency Department: a Randomized Study
Brief Title: Diagnostic Value of Portable Ultrasound for Dyspneic Patient Support in the Emergency Department
Acronym: VSCAN-DYSP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion curve too slow.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2012/XB-01; 2013-A00100-45 (Other: RCB number)
Record Dates: First submitted 2013-03-23; First posted 2013-03-27 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Dyspnea
Keywords: Vscan; portable ultrasound; emergency care; emergency room
MeSH Terms: conditions — Dyspnea; Emergencies | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Patients randomized to this arm will receive standard care.
  Intervention: Standard care.
  Interventions: Other: Standard care
- Standard care + ultrasound (Experimental): Patients randomized to this arm will receive standard care + pleuropulmonary ultrasound.
  Intervention: Standard care + ultrasound
  Interventions: Other: Standard care; Device: Vscan portable ultrasound device (GE Healthcare, Wauwatosa, WI)

INTERVENTIONS:
Other: Standard care — Standard care for dyspneic patients including contextual analysis, conventional clinical exam and a chest X-Ray.
Device: Vscan portable ultrasound device (GE Healthcare, Wauwatosa, WI) — Standard care (as described for the other intervention) + pleuropulmonary ultrasound using the Vscan portable ultrasound device (GE Healthcare, Wauwatosa, WI).
  Arms: Standard care + ultrasound

SUMMARY:
The main objective of our study is to compare the effects of two care strategies for dyspneic patients on the length of hospital stay: (1) standard care (=contextual analysis + conventional clinical chest radiography) versus (2) standard care + pleuropulmonary ultrasound.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess the following for both arms:

A-fatality rate, B-degree of concordance between the diagnosis orientation in the emergency department and final diagnosis determined by an expert committee using patient records one month later (blind evaluation by a panel of experts) C-clinical improvement between early emergency care and later care outside the emergency department (clinical parameters = blood gases and other biological parameters) D-imaging parameters.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient consulting in the emergency department for dyspnea

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient cannot read French
* The patient is pregnant, parturient, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay in days | 1 month

SECONDARY OUTCOMES:
Patient deceased? yes/no | 1 month
Diagnosis in the emergency room | upon discharge from the emergency department (max 1 month)
Diagnosis given by expert committee based on patient file | 1 month
Glasgow scale | Baseline, day 0
Glasgow scale | day 3
Heart rate | baseline, day 0
Heart rate | day 3
Respiratory rate | baseline, day 0
Respiratory rate | day 3
Systolic blood pressure | baseline, day 0
Systolic blood pressure | day 3
Diastolic blood pressure | baseline, day 0
Diastolic blood pressure | day 3
Temperature | baseline, day 0
Temperature | day 3
blood pH | baseline, day 0
blood pH | day 3
CO2 arterial pressure | baseline, day 0
CO2 arterial pressure | day 3
O2 arterial pressure | baseline, day 0
O2 arterial pressure | day 3
O2 saturation | baseline, day 0
O2 saturation | day 3
Alkaline reserve | baseline, day 0
Alkaline reserve | day 3
white blood cell count | baseline, day 0
white blood cell count | day 3
C-reactive protein | baseline, day 0
C-reactive protein | day 3
Brain Natriuretic Peptide | baseline, day 0
Brain Natriuretic Peptide | day 3
hemoglobin | baseline, day 0
hemoglobin | day 3
Pulmonary x-ray, yes/no | baseline, day 0
right alveolar opacities on x-ray, yes/no | baseline, day 0
left alveolar opacities on x-ray, yes/no | baseline, day 0
right parenchymal origin on x-ray, yes/no | baseline, day 0
left parenchymal origin on x-ray, yes/no | baseline, day 0
right pleural effusion on x-ray, yes/no | baseline, day 0
left pleural effusion on x-ray, yes/no | baseline, day 0
pleuropulmonary ultrasound, yes/no | baseline, day 0
right alveolar-interstitial syndrome on ultrasound, yes/no | baseline, day 0
left alveolar-interstitial syndrome on ultrasound, yes/no | baseline, day 0
right lung consolidation on ultrasound, yes/no | baseline, day 0
left lung consolidation on ultrasound, yes/no | baseline, day 0
right pleural effusion on ultrasound, yes/no | baseline, day 0
left pleural effusion on ultrasound, yes/no | baseline, day 0
right pneumothorax on ultrasound, yes/no | baseline, day 0
left pneumothorax on ultrasound, yes/no | baseline, day 0

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bobbia, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France